CLINICAL TRIAL: NCT05866042
Title: Boosting Psychotherapy Effects by Means of Transcranial Direct Current Stimulation
Acronym: PSYCHOBOOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PSYCHOBOOST
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2021-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active tDCS (Experimental): Administration of active tDCS, not followed by MCT session, but by a usual visit psychiatric follow-up
  Interventions: Device: tDCS
- sham tDCS and MCT (No Intervention): Administration of sham tDCS, followed by MCT session
- active tDCS and MCT (Experimental): Administration of active tDCS, followed by MCT session
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — TDCS is a noninvasive neurostimulation technique involving the transcranial application of a low-amperage electric current at a region of the cerebral cortex involved in the pathogenesis of major depression, the dorsolateral prefrontal cortex. In healthy subjects, the administration of excitatory tDCS on the left DLPFC improves the regulation of attention on information characterized by negative emotions, as does the administration of inhibitory tDCS on the DLPFC Right tDCS produces small changes in the neuronal membrane potential, thus increasing or decreasing the excitability of the stimulated tissue. Simultaneous administration to behavioral tasks designed to activate the stimulated cortical region should achieve a synergistic, amplifying the plasticity stimulated by the task.
  Arms: Active tDCS; active tDCS and MCT

SUMMARY:
The present study involves the administration of three types of interventions in patients with depressive episode in the context of DDM. Two-thirds of the patients will carry out a course of excitatory tDCS sessions on the left DLPFC, so as to improve attention regulation on information characterized by negative emotions and have an antidepressant effect, simultaneously with the performance of a task, the attentional training technique (ATT), aimed at achieve effective management of emotions characterized by negative emotions and which constitutes a fundamental exercise of MCT. In half of the patients who will undergo tDCS treatment, after each session of stimulation, an MCT session will be carried out. In addition, before and after the cycle of tDCS sessions and MCT sessions will be explored, in a subgroup of patients, in the context of a pilot study, the TMS- EEG of the change in depressive symptomatology, which can be correlated with the different proposed therapeutic interventions.

DETAILED DESCRIPTION:
The study - interventional, nonpharmacological, using medical devices, nonprofit - is aimed at evaluating the potential effectiveness of a multimodal intervention for the treatment of unipolar depression. The intervention involves the use of a neuro-stimulation technique, the Transcranial Direct Current Stimulation (transcranial Direct Current Stimulation - tDCS), combined with a psychotherapy intervention, metacognitive therapy (MetaCognitive Therapy, MCT). TDCS is a noninvasive neurostimulation technique involving the transcranial application of a low-amperage electric current at a region of the cerebral cortex involved in the pathogenesis of major depression, the dorsolateral prefrontal cortex. It has been demonstrated how such stimulation has a neuromodulating effect on synaptic plasticity, with efficacy in unipolar major depression. The technique also has a good safety, as it is not associated with major side effects. MCT is based on the metacognitive model, according to which psychopathological processes are consequent to a cognitive style characterized by repetitive forms of thinking (such as rumination) and maladaptive behaviors such as avoidance and thought suppression. The MCT, through attention training techniques, detached mindfulness and behavioral interventions on metacognitions, has shown effectiveness in major depressive disorder comparable to that of psychotherapeutic interventions considered, within psychotherapies, to be first-line such as cognitive-behavioral therapy. The experimental design will be that of a randomized, double-blind study with three arms of treatment, each consisting of 8 sessions, involving the administration of 1) the neurostimulation intervention (tDCS), 2) of the psychotherapeutic intervention alone (MCT), 3) of both techniques in consecution (tDCS-MCT). This design is aimed at evaluating a potential additive/synergistic effect of the two interventions when combined. During the tDCS sessions, each lasting 20 minutes, the patient will apply the technique of attention training, aimed at further activating the region stimulated by neurostimulation, so as to so as to amplify the plasticity stimulated by tDCS, achieving a synergistic effect. To follow, a 40-minute MCT session will be carried out. The effectiveness of these interventions will be assessed by heteroadministered and self-administered at time zero, after treatment, at two follow-ups of 6 and 12 months. Before and after the treatment cycle (tDCS sessions and MCT sessions), a subgroup of patients will be explored, in the context of a pilot study, the TMS-EEG correlates of the change in symptomatology depression, which can be correlated with the different proposed therapeutic interventions.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent to study
* Ability to understand and speak the Italian language
* DSM-5 diagnosis of Major Depressive Disorder.
* Ongoing depressive episode of at least moderate intensity (HAM-D> 18)

Exclusion Criteria:

* Previous tDCS sessions with significant side effects
* Positive personal history for seizures
* Positive family history for epileptic disease
* Positive personal history for neurological disease
* Positive personal history for head trauma with loss of consciousness
* Positive personal history for frequent and severe headaches
* Positive personal history for neurosurgical procedures
* Prior implantation of neurostimulation implants (DBS, VNS, etc.)
* Prior implantation of defibrillator or pace-maker
* Possibility of pregnancy or established pregnancy
* Substance or alcohol abuse in the past 6 months
* Positive personal history for schizophrenia or schizoaffective disorder
* Positive personal history of intellectual disability ("mental retardation")
* Current hospitalization
* Cardiac, respiratory, renal, hepatic failure, immunosuppression status

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
to evaluate the potential superiority, from the point of view of therapeutic efficacy in depression, of the approach of combined administration of tDCS and MCT, compared with interventions based tDCS alone or MCT alone. | end of treatment, 1, 3, 6 and 12 months
  Change in the Hamilton Depression Rating Scale will be used as parameters, during follow-up (end of treatment, 1, 3, 6 and 12 months).

SECONDARY OUTCOMES:
To evaluate the TMS-EEG correlates of change in depressive symptomatology, correlating them with the different proposed therapeutic interventions, in a subgroup of patients recruited, in the context of a pilot study. | 12 months
  Change, at the end of treatment, in TMS-EEG connectivity measures, in a subgroup of patients recruited 2. Change, during follow-up (end of treatment, 1, 3, 6 and 12 months), in the scores of the following scales:
  * Beck Depression Inventory
  * SCL-90
  Remorse Rating Scales:
  * Penn State Worry Questionnaire
  * Metacognition Questionnaire-30
  * Ruminative Response Scale
  * Anger rumination scale Neuropsychological tests
  * Digit span forward and backward
  * Phonemic and semantic verbal fluency

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, MI, Italy